CLINICAL TRIAL: NCT01057030
Title: Randomized, Double-Blinded, Placebo-Controlled, Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-708163 125 mg in Healthy Japanese and Non-Japanese Subjects
Brief Title: Multiple Dose Japanese Bridging Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: CN156-038
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — BMS 708163

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A1 (BMS-708163) (Active Comparator): Healthy Japanese Subjects
  Interventions: Drug: BMS-708163
- A2 (Placebo) (Placebo Comparator): Healthy Japanese Subjects
  Interventions: Drug: Placebo
- B1 (BMS-708163) (Active Comparator): Healthy Non-Japanese Subjects
  Interventions: Drug: BMS-708163
- B2 (Placebo) (Placebo Comparator): Healthy Non-Japanese Subjects
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-708163 — Capsules, Oral, 125 mg, once daily, 14 days
  Other Names: (GAMMA SECRETASE inhibitor)
  Arms: A1 (BMS-708163); B1 (BMS-708163)
Drug: Placebo — Capsules, Oral, 0 mg, once daily, 14 days
  Arms: A2 (Placebo); B2 (Placebo)

SUMMARY:
The purpose of this study is to assess the safety and tolerability of multiple oral daily doses of BMS-708163 in healthy young male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese and non-Japanese subjects
* Japanese subjects must be first generation Japanese and must demonstrate both maternal and paternal Japanese ancestry
* Non-Japanese subjects must not be of Japanese or Asian descent, ie, neither parent nor grandparent was born in Japan or in any Asian country
* BMI of 19 to 25 kg/m², for Japanese and non-Japanese subjects
* Men ages 20 to 45 years

Exclusion Criteria:

* Serum creatinine values above the normal range
* Urine protein or blood levels above the normal range
* Liver function tests above the normal range
* TSH, free T3, or free T4 outside the normal range
* Amylase or lipase levels above the normal range
* Positive Fecal Immunochemical Test (FIT™)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
BMS-708163 or placebo in Japanese and non-Japanese: Safety and tolerability (AE's, ECG, vital signs, safety labs) | Every day for 28 days

SECONDARY OUTCOMES:
BMS-708163 pharmacokinetic parameters (Cmax, Cmin, Ctrough, Tmax, AUC(TAU), AI, and CLT/F and T-HALF (only following Day 14 dose)) | Days 1, 7, and 14

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx